CLINICAL TRIAL: NCT07012213
Title: Effect of Nasal Dexmedetomidine Versus Systemic Infusion Dexmedetomidine in Reducing Intraoperative Opioid Consumption in Nasal Endoscopic Surgeries: A Prospective Randomized Controlled Study
Brief Title: Nasal Dexmedetomidine Versus Systemic Infusion Dexmedetomidine in Reducing Intraoperative Opioid Consumption in Nasal Endoscopic Surgeries
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marianne Magdy Youssef, Lecturer of anesthesia ,icu&pain management, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ms-405-2024
Record Dates: First submitted 2025-05-23; First posted 2025-06-10 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Functional Endoscopic Sinus Surgery (FESS)

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Dexmedetomidine IV infusion (0.5 mcg/kg/h) after induction (Active Comparator)
  Interventions: Drug: Patients in group A received .5 g/kg/h dexmedetomidine infusion after general anesthesia, in group B received 1 ml (100 mic) dexmedetomidine intranasal spray before induction.
- Group B: Intranasal dexmedetomidine 1 ml (100 mcg) preoperatively. (Active Comparator)
  Interventions: Drug: Patients in group A received .5 g/kg/h dexmedetomidine infusion after general anesthesia, in group B received 1 ml (100 mic) dexmedetomidine intranasal spray before induction.

INTERVENTIONS:
Drug: Patients in group A received .5 g/kg/h dexmedetomidine infusion after general anesthesia, in group B received 1 ml (100 mic) dexmedetomidine intranasal spray before induction. — Patients in group A received .5 g/kg/h dexmedetomidine infusion after general anesthesia, in group B received 1 ml (100 mic) dexmedetomidine intranasal spray before induction.

SUMMARY:
Background: Optimizing intraoperative hemodynamics and minimizing opioid use are crucial in nasal endoscopic surgeries.

Objective: To compare the efficacy of intranasal dexmedetomidine spray and intravenous dexmedetomidine infusion in reducing intraoperative opioid requirements and improving perioperative outcomes.

Methods: A prospective randomized controlled study was conducted on 50 patients undergoing nasal endoscopic surgeries. Patients will be randomized into two groups: Group A received IV dexmedetomidine infusion; Group B received intranasal dexmedetomidine. Intraoperative fentanyl use, postoperative morphine consumption, hemodynamic parameters, and pain scores will be evaluated.

Measurements:

All the following data will be collected:

* Demographic data: age, sex, weight, height, BMI, ASA class, indication and duration of surgery.
* Hemodynamic Parameters: HR, BP, SpO2, and MAP will be recorded preoperative, and every 10 min till the end of surgery.
* Quality of surgical field through endoscopic surgical field grading system Primary outcome is Reducing opioid consumption intraoperatively to give the best surgical field control and hemodynamic control. Secondary outcomes are pain score postoperative, postoperative analgesics, and surgical field satisfaction.

Statistical analysis Statistical analysis will be done by SPSS v26 (IBM Inc., Chicago, IL, USA). Shapiro-Wilks test and histograms will be used to evaluate the normality of the distribution of data. Quantitative parametric variables will be presented as mean and standard deviation (SD) and compare between the two groups utilizing unpaired Student's T- test. Quantitative non-parametric data will be presented as median and interquartile range (IQR) and will be analyzed by Mann Whitney-test. Qualitative variables will be presented as frequency and percentage (%) and will be analyzed utilizing the Chi-square test or Fisher's exact test when appropriate. A two tailed P value < 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:• Age ≥ 18 years.

* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-II.
* Patients underwent nasal endoscopic surgeries under general anesthesia.

Exclusion Criteria:• Patient refusal.

* Severe complication with the injection of dexmedetomidine as first degree or second-degree atrioventricular block, atrial fibrillation.
* Hypersensitivity to the drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2025-11-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary: Intraoperative fentanyl use. | 40 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Kasralaini medical school, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD sharing was not included in the informed consent process & there are institutional limitations on sharing individuals level data